CLINICAL TRIAL: NCT02962024
Title: Does Local Morphine Add to Local Anesthetics in Serratus Anterior Plane Block for Post Mastectomy Pain Has a System Analgesic Effect? A Clinical and Pharmacokinetics Study
Brief Title: Does Local Morphine Add to Local Anesthetics in Serratus Anterior Plane Block Has a System Analgesic Effect?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Adel El sherif,MD (Other)
Responsible Party: Sponsor-Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia, ICU and pain management, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 348
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- morphine sulphate (Active Comparator): 10mg locally morphine hydrochloride once betwwen serratus muscle and latissmus dorsi muscle
  Interventions: Drug: Morphine Sulfate
- bupivacaine hydrochloride (Placebo Comparator): 0.25%locally bupivacaine hydrochloride once
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Morphine Sulfate
  Other Names: morphine
  Arms: morphine sulphate
Drug: Bupivacaine Hydrochloride
  Other Names: marcaine
  Arms: bupivacaine hydrochloride

SUMMARY:
the investigators aim is to investigate and explore the effect 10 mg morphine added to local anesthetics in serratus anterior plane block for post mastectomy pain management after modified radical mastectomy in patients with breast cancer with assessment of its serum level if it will be absorbed systemically or not?

ELIGIBILITY:
Inclusion Criteria:

* (ASA) class I-II
* body weight of 50 - 90 kg

Exclusion Criteria:

* a history of bleeding diathesis,
* relevant drug allergy, opioid dependence,
* sepsis, prior surgery in the supraclavicular, infraclavicular or axillary regions, alcohol or drug abuse , patients with advanced cardiovascular disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
serum morphine level after local injection | 24 hours
  concentration of serum morphine in ng/ml after local injection

CONTACTS AND LOCATIONS:
Overall Officials: fatma EL sherif, Study Director — South Egypt Cancer Instuite, Assuit, Assuit university
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Sherif FA, Abd El-Rahman AM, Othman AH, Shouman SA, Omran MM, Hassan NA, Hassan SB, Aboeleuon E. Analgesic Effect of Morphine Added to Bupivacaine in Serratus Anterior Plane Block Following Modified Radical Mastectomy. Only a Local Effect? Randomized Clinical Trial. J Pain Res. 2020 Mar 31;13:661-668. doi: 10.2147/JPR.S236336. eCollection 2020. PMID 32280268